CLINICAL TRIAL: NCT06387069
Title: A Multicenter, Randomized, Open-Label, Phase III Clinical Study to Evaluate the Efficacy and Safety of HMPL-306 vs. Salvage Chemotherapy Regimens in Patients With IDH1- and IDH2-mutated Relapsed/Refractory Acute Myeloid Leukemia (R/R AML)
Brief Title: A Study to Evaluate HMPL-306 in Patients With IDH1or IDH2-mutated Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-306-00CH1
Record Dates: First submitted 2024-04-16; First posted 2024-04-26 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; IDH
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HMPL-306 arm (Experimental): HMPL-306
  Interventions: Drug: HMPL-306 Regimen
- Salvage treatment arm (Active Comparator): Salvage treatment
  Interventions: Drug: Salvage Chemotherapy Regimen

INTERVENTIONS:
Drug: HMPL-306 Regimen — Patients will receive HMPL-306 monotherapy: HMPL-306 PO at 250 mg QD (C1) + 150 mg QD (starting from C2), 28 days as a cycle.
  Arms: HMPL-306 arm
Drug: Salvage Chemotherapy Regimen — Patients in this regimen will receive treatment with one of the following regimens, and the regimen will be selected by the investigator based on the patient's condition:
  * EA±Mitox regimen: etoposide injection 100 mg/m2, cytarabine injection 100-150 mg/m2, mitoxantrone injection 8 mg/m2 QD IV for 5 consecutive days (Days 1-5).
  * FLAG ± Ida regimen: G-CSF injection 300 mcg/m2 QD SC for 5 consecutive days (Days 1-5); fludarabine injection 30 mg/m2 QD IV for 5 consecutive days (Days 2-6); cytarabine injection 1000-2000 mg/m2 QD IV for 5 consecutive days (Days 2-6); idarubicin injection 10 mg/m2 QD IV for 3 consecutive days (Days 2-4).
  * LoDAC: -Cytarabine Injection 20 mg every 12 hours, subcutaneous or IV for 10 consecutive days (Days 1-10).
  * Azacitidine: Azacitidine Injection 75 mg/m2, QD, subcutaneous or IV for 7 consecutive days (Days 1-7).
  Arms: Salvage treatment arm

SUMMARY:
This study is a multicenter, randomized, open-label, phase III clinical study (RAPHAEL) to evaluate the efficacy, safety, and PK of HMPL-306 versus salvage chemotherapy in patients with R/R AML harboring IDH1 and IDH2 mutations.

DETAILED DESCRIPTION:
Study Overview This is a multicenter, randomized, open-label, phase III clinical study to evaluate the efficacy, safety, and PK of HMPL-306 versus salvage chemotherapy in patients with IDH1- and IDH2-mutated R/R AML (RAPHAEL).

The study is open-label, and all patients will be screened centrally to determine their IDH mutation status, and based on the screening results, the patients will be assigned to the corresponding IDH1 and IDH2 cohorts of this registration study. Patients with both IDH1 and IDH2 mutations be assigned to the IDH2 cohort. The study consists of divided into two cohorts. Patients with R/R AML harboring IDH1-R132 mutation will be included in Cohort 1, and patients with R/R AML harboring IDH2-R140, R172 mutations will be included in Cohort 2. The two cohorts will be designed independently, analyzed separately, and subjected to statistical hypothesis testing separately. Patients in both cohorts will be randomly assigned according to the central randomization system (IWRS) in a 1:1 ratio into the experimental group and the control group. Patients in the experimental group will receive HMPL-306 monotherapy at the following dose: 250 mg once daily (QD) (first cycle, C1) + 150 mg QD [starting from the second cycle (C2)]; patients in the control group will receive salvage chemotherapy (1 of 4), including 4 different treatment regimens: Two intensive regimens (EA± Mitox regimen and FLAG ± Ida regimen) and two non-intensive regimens (azacitidine and LoDAC). Prior to randomization, the investigator will pre-select a salvage chemotherapy regimen based on the patient's condition, and randomization will be stratified according to patients' response to prior first-line therapy (relapse within 6 months after allogeneic HSCT, relapse after 6 months after allogeneic HSCT, primary refractory without HSCT, relapse within 6 months after achieving CR/CRh without HSCT, or relapse after 6 months after achieving CR/CRh without HSCT) and the intensity of the pre-selected chemotherapy regimen (intensive chemotherapy or weak chemotherapy).

After the patients sign the pre-screening informed consent form (ICF), pre-screening (genetic testing) will be performed to determine IDH mutation status for subsequent enrollment cohort, and if a patient wants to know about RAS or FLT3 mutation status, local testing can be used to clarify the latest RAS or FLT3 hotspot mutation. Patients who meet the inclusion criteria of this study will be randomized to the experimental group or the control group to receive treatment in 28-day cycles until one of the following conditions occurs: Treatment failure [refer to the Guidelines for Clinical Development of New Drugs for Acute Myeloid Leukemia issued by the Center for Drug Evaluation (CDE)]. The definition of "treatment failure" is recommended as: Treatment failure occurs when CR or CRh/CRi is not achieved after 2 cycles of treatment per protocol using the regimens for the intensive chemotherapy group. When using the regimens for the weak chemotherapy group and the experimental group, treatment failure occurs if CR or CRh/CRi is not achieved after 4 cycles of treatment, i.e., disease progression/relapse, death, unacceptable toxicity, receiving new anti-tumor therapy, judgment by the investigator that the patient no longer obtains clinical benefit from treatment, withdrawal from the study by the patient or his/her legally acceptable representative, loss to follow-up, or end of the study occurs, whichever occurs first (The treatment duration of EA±Mitox regimen and FLAG±Ida regimen in the chemotherapy group will be adjusted according to the actual medication, and a maximum of two treatment cycles will be used).

Crossover is not allowed for patients with progressive disease in the control group and the experimental group, and patients in the control group will not be allowed to crossover to other salvage regimens.

The information on treatment groups is as follows (same for both cohorts):

The experimental group: Patients treated with HMPL-306 monotherapy:

- The dose of HMPL-306 is 250 mg QD (C1) + 150 mg QD (starting from C2), continuous, PO, in 28-day treatment cycles.

The control group: Patients treated with one of the following regimens, and the regimen will be determined by the investigator on a case-by-case basis:

* EA±Mitox regimen: Etoposide Injection 100 mg/m2, Cytarabine Injection 100-150 mg/m2, and Mitoxantrone Injection 8 mg/m2, QD, intravenous (IV) administration for 5 consecutive days (Days 1-5). (In the case that Mitoxantrone Injection is not accessible, a regimen containing mitoxantrone liposome can be used, specifically: Mitoxantrone liposome + cytarabine + etoposide regimen: Mitoxantrone liposome 24-32 mg/m2, Day 1; Cytarabine 100-200 mg/m2, Day 1 to Day 7; and Etoposide 100 mg/m2, Days 1-5). The regimen can be used with or without mitoxantrone, which can be determined by the investigator based on the actual condition of the patient.
* FLAG±Ida regimen: G-CSF Injection 300 mcg/m2, QD subcutaneous administration for 5 consecutive days (Days 1-5); Fludarabine Injection 30 mg/m2, QD IV for 5 consecutive days (Days 2-6); Cytarabine Injection 1000-2000 mg/m2, QD IV for 5 consecutive days (Days 2-6); and Idarubicin Injection 10 mg/m2, QD IV for 3 consecutive days (Days 2-4). This regimen can be used with or without Ida, which can be determined by the investigator based on the actual condition of the patient. After the end of chemotherapy administration, the investigator will determine whether it is necessary to continue the administration of G-CSF, and if necessary, retreatment with G-CSF is allowed until absolute neutrophil count (ANC) > 0.5x109/L.
* LoDAC: Cytarabine Injection 20 mg every 12 hours, subcutaneous or IV for 10 consecutive days (Days 1-10).
* Azacitidine: Azacitidine Injection 75 mg/m2, QD, subcutaneous or IV for 7 consecutive days (Days 1-7).

Study Period:

The study includes pre-screening period, screening period, treatment period and follow-up period [including end of treatment (EOT) follow-up, safety observation follow-up, EFS follow-up, and OS follow-up].

The pre-screening period is defined as the period from signing the pre-screening ICF to obtaining the IDH1 and IDH2 mutation testing reports. For patients without previous IDH1 or IDH2 testing reported, specimens should be sent to the central laboratory for IDH1 and IDH2 mutation testing and other companion gene testing after signing the pre-screening ICF and prior to screening. Patients with a previously reported positive IDH1 and/or IDH2 mutation test may proceed directly to screening without pre-screening if approved by the investigator. The results confirmed by the central laboratory are required for enrollment.

The screening period is defined as the period from signing the main screening ICF to Cycle 1 Day 1 pre-dose.

Treatment period is defined as the period from the first dose to EOT. EOT Follow-up: Patients with EOT need to return to the site for EOT follow-up within 1-7 days after discontinuing treatment, or before starting other anti-tumor therapy, whichever occurs first.

Safety Observation Follow-up: Patients with EOT need to return to the site for Safety Observation Follow-up within 30 (±7) days after the last dose of study drug treatment or before starting other anti-tumor therapy, whichever occurs first.

EFS Follow-up: Patients with EOT (except for EOT due to disease progression/relapse) will be advised to remain in the study for EFS follow-up, and patients without medication after randomization will also be advised for EFS follow-up, from the day of entering EFS follow-up, and then every 8 weeks until disease progression/relapse, death, withdrawal by the patient or his/her legally acceptable representative, patient lost to follow-up, or end of study, whichever occurs first. Subsequent new transplant conditioning regimens or new anti-tumor treatment regimens will be documented during EFS follow-up.

OS Follow-up: Patients who have been randomized and have completed EFS follow-up (and who have EOT due to disease progression/relapse) will receive OS follow-up every 8 weeks from the date they enter OS follow-up until death, withdrawal by the patient and his/her legally acceptable representative, loss to follow-up, or end of study, whichever occurs first. If a patient withdraws from treatment and not from the entire study, EFS and OS data collection will be continued.

End of Study Inconsistent time of end of study is allowed between the two cohorts. The end of study for each cohort is defined as the time when the target number of OS events for the final analysis is reached in the cohort. The actual duration of study for each cohort will depend on the actual enrollment rate, dropout rate, and the length of median OS in each group.

Efficacy Assessment(s) Efficacy evaluation will be based on modified 2022 European Leukemia Net (ELN) criteria. Efficacy assessment will be performed once for each of the first 6 cycles of study drug treatment (i.e., C2D1, C3D1, C4D1, C5D1, C6D1, C7D1) and every 2 cycles after 6 cycles of treatment (i.e., C9D1, C11D1, C13D1, ......); Efficacy assessments will also be performed at the Safety Observation Follow-up and each EFS Follow-up.

Safety Assessment(s) All adverse events (AEs) will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA). The number and incidence of treatment-emergent adverse events (TEAEs) will be summarized by system organ class and preferred term.

All the serious adverse events (SAEs) related with the study procedure will be collected from the date of the signing of informed consent form for pre-screening to the date of the signing of master informed consent form; all the SAEs will be collected from the date of the signing of master informed consent form to the date when the first dose is given; all AEs/SAEs will be collected from the date when the first dose is given to 30 days after the last dose is given, or the date when a new anti-tumor therapy is started, whichever occurs first (If HSCT is performed, safety data on and after HSCT treatment will no longer be collected; If a patient experiences disease recurrence after HSCT and is re-enrolled to receive HMPL-306 treatment, the adverse events after HSCT need to be collected); SAEs confirmed by the investigator to have a reasonable possibility of correlation with the study drug will be collected 30 days after the last dose or after the start of a new antitumor therapy, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed the ICF;
2. Be able to follow the requirements of study protocol;
3. Age ≥18 years;
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 to 2;
5. Cohort 1: Patients with R/R primary AML harboring IDH1-R132 site mutation [WHO 2022 Classification Criteria for Myeloid Neoplasms and Acute Leukemia, with the exception of APL (AML-M3) and extramedullary recurrence of leukemia alone without bone marrow involvement]; Cohort 2: Patients with R/R primary AML harboring IDH2-R140/R172 mutations [WHO 2022 Classification Criteria for Myeloid Neoplasms and Acute Leukemia, with the exception of APL (AML-M3) and recurrence of extramedullary leukemia alone without bone marrow involvement]. A patient with both IDH1 and IDH2 mutations will be included in Cohort 2 (IDH2 mutation group);
6. Agree to undergo bone marrow aspiration and/or biopsy before and during treatment;
7. Be willing to complete QoL assessments at specified time points during study treatment and after treatment discontinuation;
8. Female patients of childbearing potential must agree to use highly effective contraceptive methods during the study and within 30 days after discontinuation of the study drug (the time limit of contraception for the chemotherapy group needs to be extended to 6 months after the last dose) (see Appendix 9 (contraception requirements) for more information), and agree not to donate eggs (oocytes) for reproductive purposes during this period; patients must not be lactating and must have a negative pregnancy test (if of childbearing potential);
9. Male patients with female partners of childbearing potential must use condoms during intercourse and avoid donating or freezing sperm during the study and within 30 days after discontinuation of the study drug (the time limit of contraception for the chemotherapy group needs to be extended to 6 months after the last dose).
10. Predicted survival greater than 12 weeks as assessed by the investigator.

Exclusion Criteria:

Patients who meet any of the following criteria must be excluded:

1. Patients who received prior treatment with IDH1 inhibitors, IDH2 inhibitors, or IDH1/IDH2 dual target inhibitors;
2. Patients with known RAS or FLT3 hotspot mutations (patients who have test results definitely switched to negative at the time of enrollment can be enrolled);

   Hotspot mutations include:

   KRAS mutations: G12 or G13 (exon 2); Q61 (exon 3) NRAS mutations: G12 or G13 (exon 2); Q61 (exon 3) FLT3 mutations: ITD; TKD (D835 or I836)
3. Inadequate organ function, as defined below:

   * Serum total bilirubin (TBIL) higher than 1.5 times the upper limit of normal (ULN), excluding the following patients:

     - Patients with Gilbert's disease, with normal alanine aminotransferase (ALT) and aspartate aminotransferase (AST), and serum TBIL ≤ 3 × ULN.
   * AST or ALT > 2.5 × ULN (if leukemia invades the liver, patients with AST and ALT levels ≤ 5 × ULN can be enrolled);
   * Estimated creatinine clearance by Cockcroft-Gault formula < 50 mL/min or creatinine > 1.5 × ULN;
4. International Normalized Ratio (INR) > 1.5 × ULN or activated partial thromboplastin time (aPTT) > 1.5 × ULN, except for patients who are receiving anticoagulant therapy;
5. Blood amylase > 1.5 × ULN and assessed to be clinically significant by the investigator;
6. Current known history of liver disease, including cirrhosis, alcoholic liver disease, active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV):

   * Patients who are positive for serum hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) are required to undergo HBV deoxyribonucleic acid (DNA) testing, and patients with HBV DNA test results that are either negative or below the lower limit of normal at the site can be enrolled;
   * Patients with positive HCV serology may be enrolled only if the HCV ribonucleic acid (RNA) test is negative or below the lower limit of normal at the site;
7. Known human immunodeficiency virus (HIV) infection;
8. Meet any of the following cardiac function-related criteria:

   * Any clinically significant rhythm or conduction abnormalities requiring clinical intervention;
   * Clinically significant cardiovascular diseases that require clinical intervention as judged by the investigator, including but not limited to: acute myocardial infarction, unstable angina pectoris, coronary artery bypass grafting within 6 months prior to randomization, New York Heart Association (NYHA) Class II (inclusive) or above congestive heart failure, left ventricular ejection fraction (LVEF) < 45%, or uncontrolled hypertension after medication (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg);
   * Congenital long QT syndrome or QTcF >470 msec in females/QTcF >450 msec in males;
   * Use of drugs currently known to cause QT prolongation (Appendix 5); patients who have switched the medication by 5 half-lives of the drug prior to the dosing of the study drug or have their ECG to be regularly monitored during the study (QTcF is required to be regularly monitored if no medication is available for replacement) could be enrolled.
9. Patients with other primary malignancies within the last 5 years, except for patients who have been cured, and patients with the following non-invasive tumors who have been treated with definitive treatment:

   * Basal cell carcinoma of skin
   * Squamous cell carcinoma of skin and cervix
   * Carcinoma in situ of cervix
   * Breast cancer in situ
10. Pregnant (positive pregnancy test prior to treatment) or lactating women;
11. Patients with childbearing requirements;
12. History of stroke or intracranial hemorrhage within 6 months prior to randomization;
13. Patients who have undergone major surgery within 4 weeks prior to randomization;
14. Patients who have received any monoclonal antibody for anti-tumor therapy within 3 weeks or 2 half-lives prior to randomization, whichever is longer;
15. Patients who have received treatment with the investigational product or investigational device in a clinical study within 3 weeks prior to randomization;
16. Patients who have received anti-tumor treatment (chemotherapy, targeted therapy, immunotherapy, or anti-tumor vaccine, etc,) within 3 weeks prior to randomization or received radiotherapy within 3 months prior to randomization; patients who have received CAR-T therapy within 4 weeks prior to randomization; patients who have received HSCT within 60 days prior to randomization, or are receiving immunosuppressive therapy after HSCT at screening, or are accompanied by graft-versus-host disease (GVHD) requiring drug control; patients undergoing treatment for skin graft-versus-host disease (GVHD) with fixed oral doses of and/or topical corticosteroids may be enrolled only if they can benefit from the study treatment as assessed by the investigator; for patients receiving prophylactic intrathecal administration of chemotherapy drugs (cytarabine, dexamethasone and methotrexate) to prevent central leukemia, no washout is required;
17. Central nervous system leukemia: patients with clinical symptoms suggesting active central nervous system (CNS) leukemia or confirmed CNS leukemia invasion;
18. Patients who have received live vaccines within 4 weeks prior to randomization;
19. Use of traditional Chinese medicine with anti-tumor effect within 1 week prior to randomization;
20. Patients with uncontrolled active systemic fungal, bacterial, or viral infection (defined as persistent signs/symptoms related to the infection without improvement despite appropriate antibiotic or antiviral therapy and/or other treatments), or persistent unexplained pyrexia (> 38.5℃) without improvement during the screening period (only patients with tumor fever as judged by the investigator can be enrolled);
21. Inability to take medications orally, past surgery history or severe gastrointestinal diseases including dysphagia, active gastric ulcer, etc., which may interfere with the absorption of study drug as judged by the investigator;
22. Insufficient compliance in participating in this clinical study as judged by the investigator;
23. Toxicities from previous anti-tumor treatments have not yet recovered to Grade ≤ 1 (excluding alopecia);
24. Patients with any other disease, metabolic abnormality, physical examination abnormality or clinically significant laboratory test abnormality, based on which the investigator has reason to suspect that the patient has certain disease or condition that is not suitable for treatment with the investigational product, or that will affect the interpretation of study results or will put the patient at high risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
OS | Up to approximately 33 months
  Overall survival (OS)

SECONDARY OUTCOMES:
CR rate | Up to approximately 33 months
  Proportion of patients who achieve a complete remission (CR)
CR + CRh rate | Up to approximately 33 months
  Proportion of patients who achieve complete remission plus complete remission with partial hematologic recovery rate
CR + CRi + CRh rate | Up to approximately 33 months
  Proportion of patients who achieve complete remission plus complete remission with incomplete hematologic recovery and partial hematologic recovery rate
Assessments for PK (pharmacokinetics) | Day1 of cycle 1, 3, 5 (each cycle is 28 days)，up to approximately 33 months
  Maximum Plasma concentration (Cmax) of drug
Assessments for PK (pharmacokinetics) | Day1 of cycle 1, 3, 5 (each cycle is 28 days)，up to approximately 33 months
  Trough plasma concentration (Ctrough) of drug
Duration of response (DOR) | Up to approximately 33 months
  Duration of CR (DoCR), duration of CR + CRh, duration of CR + CRh + Cri
Transfusion-dependence conversion ratio | Up to approximately 33 months
HSCT(hematopoietic stem cell transplantation) ratio | Up to approximately 33 months
Safety（TEAE, TRAE, SAE, etc.） | Up to approximately 33 months
  Number of participants with treatment-related adverse events, treatment-emergent adverse events, serious adverse events, adverse events leading to dose modification, adverse events leading to death as assessed by CTCAE v5.0
Quality of life (QoL) | Up to approximately 33 months
  Quality of life (QoL), as measured by Family Reported Outcome Measure (Form-Item Health Survey)
Time to response (TTR) | Up to approximately 33 months
  Time to first CR (TTCR), time to first CR + CRh [TT (CR + CRh)], time to first CR + CRh + CRi [TT (CR + CRi + CRh)]
EFS | Up to approximately 33 months
  Event-free survival (EFS)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Doctor, Principal Investigator — Peking University People's Hospital
Locations (53):
- China (53):
  - Anhui Provincial Hospital（The First Affiliated Hospital of U STC）, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affilated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Quanzhou First Hospital Affiliated to Fujian Medical University, Quanzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital，Southern Medical University, Guanzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical Univercity, Zunyi, Guizhou
  - Baoding NO.1 Central Hospital, Baoding, Hebei
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin First Hospital, Harbin, Heilongjiang
  - The First Affilated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - People's Hospital of Hunan Province, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xi'an Jiaotong University (Xibei Hosiptal), Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The second people's hospital of Yibin, Yibin, Sichuan
  - XinjiangUiger Municipal People's Hospital, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of WMU, Wenzhou, Zhejiang
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin
  - Tianjin People's Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu L, Wei X, Zhao W, Hu Y, Li J, Dong Y, Gong T, Zhang X, Xu Y, Zhang Y, Xu C, Zhang C, Cai Z, Jing H, Mi R, Wu W, He W, Wang H, Tang Q, Jiang Z, Liu H, Chen G, Sun J, Chen J, Yan S, Yan H, Wangwu J, Zhong Z, Wang L, Fan S, Shi M, Su W, Huang X. HMPL-306 in relapsed or refractory IDH1- and/or IDH2-mutated acute myeloid leukemia: A phase 1 study. Med. 2025 Jun 13;6(6):100575. doi: 10.1016/j.medj.2025.100575. Epub 2025 Jan 31. PMID 39892383